CLINICAL TRIAL: NCT01470924
Title: High Curability Via Intensive Reinduction Chemotherapy and Stem Cell Transplantation in Young Adults With Relapsed Acute Lymphoblastic Leukemia in Sweden 2003-2007
Brief Title: Acute Lymphoblastic Leukemia Relapse in Sweden 2003-2007
Status: Completed | Type: Observational
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Piotr Kozlowski, Principal Investigator, Region Örebro County
Other Study IDs: OLL-180361
Record Dates: First submitted 2011-11-07; First posted 2011-11-11 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: acute lymphoblastic leukemia; relapse; salvage; prognostic
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
A minority of patients with adult acute lymphoblastic leukemia (ALL) relapse are rescued. The aim of this population-based study was to assess the results of reinduction treatment and allogeneic stem cell transplantation (SCT) in second complete remission (CR) in Sweden 2003-2007.

DETAILED DESCRIPTION:
This is a national, multicenter, prospective, population-based study of outcome among adult patients aged 19 to 65 years with ALL relapse diagnosed during 2003-2007 in Sweden. Most of the patients had primary treatment according to National guidelines for ALL as recommended by The Swedish Adult ALL Group (SVALL). The guidelines suggest two different treatment protocols for early relapses, and retreatment according to the initial therapy for late relapses, with the intention to proceed to allogeneic SCT in CR2 for eligible patients. The aim of the current study was to assess outcome among adult patients after first ALL relapse, and the utilization and efficacy of recommended protocols and of allogeneic SCT in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with first relapse of ALL

Exclusion Criteria:

* patients with Burkitt leukemia

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults with relapsed ALL
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2003-01; Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Piotr J Kozlowski, MD, Principal Investigator — Region Örebro County
Locations (1):
- Orebro University Hospital, Örebro, Örebro County, Sweden